CLINICAL TRIAL: NCT04515641
Title: An Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of Islatravir (MK-8591) in Participants With Moderate Hepatic Impairment
Brief Title: Single-Dose Islatravir in Moderate Hepatic Impairment (MK-8591-030)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8591-030; MK-8591-030 (Other: MSD)
Record Dates: First submitted 2020-08-14; First posted 2020-08-17 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Human Immunodeficiency Virus (HIV) Infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — islatravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moderate Hepatic Impairment (Experimental): Participants receive a single dose of ISL 60 mg.
  Interventions: Drug: Islatravir
- Healthy Controls (Experimental): Participants receive a single dose of ISL 60 mg.
  Interventions: Drug: Islatravir

INTERVENTIONS:
Drug: Islatravir — Two ISL 30 mg capsules taken by mouth.
  Other Names: MK-8591

SUMMARY:
This is an open-label, single-dose study of the plasma pharmacokinetics (PK), safety, and tolerability of islatravir (ISL, MK-8591), and the intracellular PK of ISL triphosphate (ISL-TP) in male and female adult participants with moderate hepatic impairment and in healthy matched control participants.

ELIGIBILITY:
Inclusion Criteria:

Healthy Control Participants:

* Is in good health based on medical history, physical examination, vital sign (VS) measurements and electrocardiograms (ECGs) performed prior to randomization
* Is in good health based on laboratory safety tests obtained at the screening visit and prior to administration of the initial dose of study drug.
* Has a body mass index (BMI) ≥18.5 and ≤40 kg/m2

Hepatic Impairment Participants:

* Has a diagnosis of chronic (> 6 months), stable (no acute episodes of illness within the previous 2 months due to deterioration in hepatic function) hepatic insufficiency with features of cirrhosis due to any etiology
* Has a score on the Child-Pugh scale ranging from 7 to 9 (moderate hepatic insufficiency) at screening
* With the exception of hepatic impairment, is in generally good health
* Has a BMI ≥ 18.5 and ≤ 40 kg/m2

Healthy and Hepatic Impairment Participants:

* Males : uses contraception according to local regulations
* Females: is not pregnant or breastfeeding and one of the following applies:
* Is not a woman of childbearing potential (WOCBP) OR
* Is a WOCBP and uses an acceptable contraceptive method
* A WOCBP with negative highly sensitive pregnancy test within 24 hours of study intervention

Exclusion Criteria:

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of clinically significant psychiatric disorder of the last 5 years
* Has a history of cancer (malignancy)
* Has a history of significant multiple and/or severe allergies, or has had an anaphylactic reaction or significant intolerability (ie, systemic allergic reaction) to prescription or non-prescription drugs or food
* Has known hypersensitivity to the active substance or any of the excipients of the study drug
* Is positive for hepatitis B surface antigen, hepatitis C antibodies, HIV-1 or HIV-2
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy (screening) visit
* Is unable to refrain from or anticipates the use of any medication, including prescription and nonprescription drugs or herbal remedies beginning approximately 2 weeks (or 5 half-lives) prior to study drug administration, throughout the study, until the poststudy visit
* Has participated in another investigational study within 4 weeks (or 5 half-lives, whichever is greater) prior to the prestudy (screening) visit
* Has a QTc interval >470 for males or >480 ms for females, has a history of risk factors for Torsades de Pointes (eg, heart failure/cardiomyopathy or family history of long QT syndrome), has uncorrected hypokalemia or hypomagnesemia, is taking concomitant medications that prolong the QT/QTc interval
* Is not considered low risk of having HIV infection
* Is a smoker or user of electronic cigarettes and/or has used nicotine or nicotine-containing products (eg, nicotine patch) within 3 months of screening
* Consumes greater than 3 glasses of alcoholic beverages per day
* Consumes more than 6 caffeinated beverages per day
* Is a regular user of illicit drugs or has a history of drug abuse within 2 years
* Presents any concern to the investigator regarding safe study participation
* Is unwilling to comply with study restrictions
* Is or has an immediate family member who is investigational site or Sponsor staff directly involved with this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Clinical Pharmacology of Miami ( Site 0001), Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Matthews RP, Patel M, Liu W, Liu Y, Rondon JC, Vargo RC, Stoch SA, Iwamoto M. Pharmacokinetics of islatravir in participants with moderate hepatic impairment. Antimicrob Agents Chemother. 2025 Apr 2;69(4):e0155324. doi: 10.1128/aac.01553-24. Epub 2025 Mar 5. PMID 40042304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and females with moderate hepatic impairment between the ages of 18 and 75 years old (inclusive), and healthy matched controls were enrolled in this study
Groups:
- Participants With Moderate Hepatic Impairment: Participants with moderate hepatic impairment received a single oral dose of 60 mg Islatravir administered in capsule form.
- Healthy Matched Control Participants: Healthy participants received a single oral dose of 60 mg Islatravir administered in capsule form.
Period: Overall Study
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (9.4) | 59.5 (6.6) | 60.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time 0 to Infinity (AUC0-inf) of Islatravir (ISL) in Plasma
Description: Participants were treated with ISL, and blood samples were collected from pre-dose up to 168 hours post-dose to determine the concentration of plasma ISL. The 95% confidence interval was derived from a fixed effects model performed on natural log-transformed values.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 168 hours post-dose
Population: Participants who comply with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance covers such considerations as exposure to treatment, availability of measurements and absence of important protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: Hours*μmol/Liter
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Number analyzed (Participants) | 6 | 6
Hours*μmol/Liter | 5.81 [5.08 to 6.64] | 7.74 [5.67 to 10.6]
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Impairment vs Healthy Matched Control Participants; Geometric least-squares mean ratio (GMR); Test type: Other; GMR = 0.75, 90% CI 2-sided [0.58 to 0.96] — Participants with Moderate Hepatic Impairment / Healthy Matched Control Participants; GMR calculated using the mean square error referencing a t-distribution. Confidence limits exponentiated to obtain the 90% confidence interval

2. Primary Outcome: Area Under the Curve From Time 0 to Last Sampling Time (AUC0-last) of ISL in Plasma
Description: as for outcome 1
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Hours*μmol/Liter
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Number analyzed (Participants) | 6 | 6
Hours*μmol/Liter | 5.25 [4.55 to 6.07] | 6.97 [5.04 to 9.63]
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Impairment vs Healthy Matched Control Participants; Geometric least-squares mean ratio (GMR); Test type: Other; GMR = 0.75, 90% CI 2-sided [0.58 to 0.98] — Participants with Moderate Hepatic Impairment / Healthy Matched Control Participants; [other analysis details as in outcome 1, analysis 1]

3. Primary Outcome: Maximum Concentration (Cmax) of ISL in Plasma
Description: as for outcome 1
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μmol/Liter
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Number analyzed (Participants) | 6 | 6
μmol/Liter | 0.834 [0.440 to 1.58] | 1.28 [0.822 to 1.98]
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Impairment vs Healthy Matched Control Participants; Geometric least-squares mean ratio (GMR); Test type: Other; GMR = 0.65, 90% CI 2-sided [0.38 to 1.14] — Participants with Moderate Hepatic Impairment / Healthy Matched Control Participants; [other analysis details as in outcome 1, analysis 1]

4. Primary Outcome: Time to Maximum Concentration (Tmax) of ISL in Plasma
Description: Participants were treated with ISL, and blood samples were collected from pre-dose up to 168 hours post-dose to determine the concentration of plasma ISL. The Tmax of plasma ISL was expressed as a median.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 168 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Number analyzed (Participants) | 6 | 6
Hours | 1.00 [1.00 to 6.00] | 1.00 [1.00 to 2.00]

5. Primary Outcome: Apparent Terminal Half-Life (t½) of ISL in Plasma
Description: Participants were treated with ISL, and blood samples were collected from pre-dose up to 168 hours post-dose to determine the concentration of plasma ISL. The Geometric Coefficient of Variation was expressed as a percent (%CV), and is calculated from the square root of corresponding estimated variance obtained for each population in fixed effect model multiplied by 100.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Number analyzed (Participants) | 6 | 6
Hours | 72.9 (13.6) | 83.9 (12.0)

6. Primary Outcome: Apparent Total Clearance (CL/F) of ISL in Plasma
Description: as for outcome 5
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/Hour
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Number analyzed (Participants) | 6 | 6
Liters/Hour | 35.1 (12.9) | 26.5 (30.3)

7. Primary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/F) of ISL in Plasma
Description: as for outcome 5
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, and 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Number analyzed (Participants) | 6 | 6
Liters | 3714 (18.4) | 3197 (38.6)

8. Secondary Outcome: Percentage of Participants With an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Time Frame: Up to 28 days
Population: All participants who received at least one dose of treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Number analyzed (Participants) | 6 | 6
Percentage of participants | 16.7 | 16.7

9. Secondary Outcome: Percentage of Participants Who Discontinued From the Study Due to an AE
Description: as for outcome 8
Time Frame: Up to 28 days
Population: All participants who received at least one dose of treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Number analyzed (Participants) | 6 | 6
Percentage of participants | 0.0 | 0.0

10. Secondary Outcome: AUC0-inf of ISL Triphosphate (ISL-TP) in Peripheral Blood Mononuclear Cells (PBMC)
Description: Participants were treated with ISL, and peripheral blood samples were collected from pre-dose up to 672 hours post-dose to determine the concentration of ISL-TP in PBMCs. The 95% confidence interval was derived from a fixed effects model performed on natural log-transformed values.
Time Frame: Predose and 4, 24, 48, 96, 168, 240, 336, 408, 504, and 672 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hours*μmol/Liter
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Number analyzed (Participants) | 6 | 6
hours*μmol/Liter | 19500 [15200 to 25000] | 25700 [19000 to 34700]
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Impairment vs Healthy Matched Control Participants; Geometric least-squares mean ratio (GMR); Test type: Other; GMR = 0.76, 90% CI 2-sided [0.57 to 1.00] — Participants with Moderate Hepatic Impairment / Healthy Matched Control Participants; [other analysis details as in outcome 1, analysis 1]

11. Secondary Outcome: AUC0-last of ISL-TP in PBMC
Description: Participants were treated with ISL and peripheral blood samples were collected from pre-dose up to 672 hours post-dose to determine the concentration of ISL-TP in PBMCs. The 95% confidence interval was derived from a fixed effects model performed on natural log-transformed values.
Time Frame: Predose and 4, 24, 48, 96, 168, 240, 336, 408, 504, and 672 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hours*μmol/Liter
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Number analyzed (Participants) | 6 | 6
hours*μmol/Liter | 18600 [14700 to 23500] | 24100 [17300 to 33600]
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Impairment vs Healthy Matched Control Participants; Geometric least-squares mean ratio (GMR); Test type: Other; GMR = 0.77, 90% CI 2-sided [0.58 to 1.03] — Participants with Moderate Hepatic Impairment / Healthy Matched Control Participants; [other analysis details as in outcome 1, analysis 1]

12. Secondary Outcome: Cmax of ISL-TP in PBMC
Description: as for outcome 11
Time Frame: Predose and 4, 24, 48, 96, 168, 240, 336, 408, 504, and 672 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μmol/Liter
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Number analyzed (Participants) | 6 | 6
μmol/Liter | 109 [83.7 to 141] | 113 [68.0 to 189]
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Impairment vs Healthy Matched Control Participants; Geometric least-squares mean ratio (GMR); Test type: Other; GMR = 0.96, 90% CI 2-sided [0.63 to 1.46] — Participants with Moderate Hepatic Impairment / Healthy Matched Control Participants; [other analysis details as in outcome 1, analysis 1]

13. Secondary Outcome: Concentration at 24 Hours Post Dose (C24) of ISL-TP in PBMC
Description: Participants were treated with ISL and peripheral blood samples were collected at 24 hours post-dose to determine the concentration of ISL-TP in PBMCs. The 95% confidence interval was derived from a fixed effects model performed on natural log-transformed values.
Time Frame: 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μmol/Liter
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Number analyzed (Participants) | 6 | 6
μmol/Liter | 103 [74.7 to 141] | 97.6 [54.3 to 175]
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Impairment vs Healthy Matched Control Participants; Geometric least-squares mean ratio (GMR); Test type: Other; GMR = 1.05, 90% CI 2-sided [0.65 to 1.71] — Participants with Moderate Hepatic Impairment / Healthy Matched Control Participants; [other analysis details as in outcome 1, analysis 1]

14. Secondary Outcome: Concentration at 168 Hours Post Dose (C168) of ISL-TP in PBMC
Description: Participants were treated with ISL and peripheral blood samples were collected at 168 hours post-dose to determine the concentration of ISL-TP in PBMCs. The 95% confidence interval was derived from a fixed effects model performed on natural log-transformed values.
Time Frame: 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μmol/Liter
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Number analyzed (Participants) | 6 | 6
μmol/Liter | 39.9 [30.0 to 53.1] | 46.4 [29.6 to 72.6]
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Impairment vs Healthy Matched Control Participants; Geometric least-squares mean ratio (GMR); Test type: Other; GMR = 0.86, 90% CI 2-sided [0.59 to 1.26] — Participants with Moderate Hepatic Impairment / Healthy Matched Control Participants; [other analysis details as in outcome 1, analysis 1]

15. Secondary Outcome: Concentration at 672 Hours Post Dose (C672) of ISL-TP in PBMC
Description: Participants were treated with ISL and peripheral blood samples were collected at 672 hours post-dose to determine the concentration of ISL-TP in PBMCs. The 95% confidence interval was derived from a fixed effects model performed on natural log-transformed values.
Time Frame: 672 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μmol/Liter
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Number analyzed (Participants) | 6 | 6
μmol/Liter | 3.80 [2.25 to 6.42] | 5.82 [4.38 to 7.74]
Statistical Analysis 1: Comparison: Participants With Moderate Hepatic Impairment vs Healthy Matched Control Participants; Geometric least-squares mean ratio (GMR); Test type: Other; GMR = 0.65, 90% CI 2-sided [0.42 to 1.01] — Participants with Moderate Hepatic Impairment / Healthy Matched Control Participants; [other analysis details as in outcome 1, analysis 1]

16. Secondary Outcome: Tmax of ISL-TP in PBMC
Description: Participants were treated with ISL and peripheral blood samples were collected from pre-dose up to 672 hours post-dose to determine the concentration of ISL-TP in PBMCs. The Tmax of ISL-TP was expressed as a median.
Time Frame: Predose and 4, 24, 48, 96, 168, 240, 336, 408, 504, and 672 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Number analyzed (Participants) | 6 | 6
Hours | 24.00 [4.00 to 48.00] | 48.00 [24.00 to 96.00]

17. Secondary Outcome: T1/2 of ISL-TP in PBMC
Description: Participants were treated with ISL, and peripheral blood samples were collected from pre-dose to 672 hours post-dose to determine the concentration of ISL-TP in PBMCs. The Geometric Coefficient of Variation was expressed as a percent (%CV), and is calculated from the square root of corresponding estimated variance obtained for each population in fixed effect model multiplied by 100.
Time Frame: Predose and 4, 24, 48, 96, 168, 240, 336, 408, 504, and 672 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
Number analyzed (Participants) | 6 | 6
Hours | 148 (18.4) | 169 (31.9)

ADVERSE EVENTS:
Time Frame: Up to 28 days
Description: All-cause mortality includes all allocated participants and safety includes all participants who received at least one dose of study treatment.
Arm/Group | Participants With Moderate Hepatic Impairment | Healthy Matched Control Participants
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Moderate Hepatic Impairment (N=6) | Healthy Matched Control Participants (N=6)
Headache (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/41/NCT04515641/Prot_SAP_000.pdf